CLINICAL TRIAL: NCT06683027
Title: Nonattachment Training for Post Traumatic Stress Recovery: a Pilot Randomised Controlled Trial
Brief Title: Nonattachment Training for Post Traumatic Stress Recovery
Acronym: NPTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Derby (Other)
Responsible Party: Principal Investigator, Lindsay Tremblay, Principal Investigator, University of Derby
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ETH2425-0417
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Post Traumatic Stress Symptoms; PTSD
Keywords: nonattachment; post traumatic stress; co-creation; NPTS; nonattachment for post traumatic stress; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: There are two conditions.
  1: Experimental group receives access to the online intervention immediately. 2. Treatment as Usual (TAU) group receives delayed (10 weeks) access to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group 1 (Experimental): This group will receive the first round of access to the program.
  Interventions: Behavioral: Nonattachment for Post Traumatic Stress
- Treatment as Usual (Active Comparator): This group will be given access to the program 10 weeks after group 1 so that data from each condition can be compared.
  Interventions: Behavioral: Nonattachment for Post Traumatic Stress

INTERVENTIONS:
Behavioral: Nonattachment for Post Traumatic Stress — This study seeks to cultivate nonattachment specifically for the alleviation of symptoms of post-traumatic stress. This is an 8-week online intervention where, following a Qualrics-hosted pre-screen, users are directed to www.npts.online to use as they wish. Users are then solicited to re-take quantitative assessments, and a subset of 10 (target number) will be recruited for a qualitative interview regarding their experience of the intervention.
  A final prompt for assessment re-takes will follow at 3 months post-intervention to determine longitudinal efficacy.

SUMMARY:
This pilot study aims to investigate the effectiveness of a novel, co-created intervention based on principles of nonattachment for individuals recovering from Post-Traumatic Stress (PTS).

Objectives include:

1. Determine whether participants undertaking nonattachment-based training have higher levels of nonattachment (as indicated by NAS Scale) after completing program.
2. Determine whether nonattachment levels are impacted after 3 months
3. Determine whether PTS symptoms are impacted by training/intervention

DETAILED DESCRIPTION:
This study will be a pilot randomised controlled trial with an embedded qualitative arm, which will be used to analyse and refine the novel intervention for a second RCT in the future. The study will be registered in a trial registry upon confirmation of ethics approval.

Recruitment will take place primarily through PTSD UK, the organisation that has generously permitted access to social media followers for the co-creation of the intervention itself (Appendix B). Recruitment points will also include Reddit, Facebook, Instagram, and threads/X sites operated by the researcher and their supervisor as well as other relevant groups (permission to post the advert will be sought from the sight admin as appropriate).

Participants will be screened for exclusionary criteria, and then, upon meeting appropriate inclusionary criteria, be prompted to undertake the following baseline assessments:

* Nonattachment Scale (NAS)- a 30-item Likert scale informed by Buddhist principles measuring aspects such as psychological flexibility, nonreactivity, and capacity for recovery after emotional disturbance.
* The Acceptance and Action Questionnaire - version II (AAQ-II) - a 7-item Likert scale measuring psychological inflexibility and experiential avoidance.
* FFMQ- a 39-item Likert scale derived from factor analysis of multiple existing assessments designed to measure mindfulness in daily life.
* Posttraumatic Stress Disorder Checklist (PCL-5) in which participants are prompted to rate on a 5-point Likert scale how much each of the 20 included problems or complaints.
* International Trauma Questionnaire (ITQ) - an 18-item Likert scale based on the World Health Organisation's ICD-11 principles for PTSD and CPTSD.

These assessments (except for NAS) were commonly utilised in the systematic review of nonattachment in clinical applications.

Following these assessments, users can access an online version of the NPTS intervention.

Pre-screening will be hosted by Qualtrics for data security, and the course itself will be hosted by Squarespace, a fully GDPR compliant platform, which also permits the researcher access to analytics to ensure participants have actually completed the course content, and to analyse for data related to module popularity and user feedback. There are 8 modules, which can be completed in any order, on the preferred schedule of the user. The user will be informed that they have 8 weeks to complete the program, after which time their data will not be included in the analysis if they have not completed the program. Each module could take as little as 10 minutes, or as long as an hour depending on the pace and depth at which the user chooses to engage with the content. Following the 8-week open access, the user will be thanked for their participation, and will be asked to re-take the assessments taken at baseline to determine intervention impact.

GDPR Compliance and data privacy and protection features of Squarespace can be found here: https://support.squarespace.com/hc/en-us/articles/360000851908-GDPR-and-Squarespace?platform=v6&websiteId=6703dafa02530b592b6006ba

However, no personal, identifiable participant information will be collected or stored on Squarespace.

Outline of study methods

Procedure:

Invitations to participate (Appendix C) will be advertised on social media platforms designed for groups who are likely to have been exposed to traumatic events or suffering from PTS-type symptoms.

Participants interested in participating will be invited to click on a link taking them to Qualtrics and the following forms:

i. Participant Information sheet informing them on what their participation entails, including the potential for delayed timing of the training to account for conditions of study design (also contained within Appendix C)

ii. Data protection and rights form (Appendix D)

iii. Consent form (Appendix E)

iv. Demographic and screening questions (Appendix F)

Participants will be asked to acknowledge their reading and understanding of this material.

Participants will be asked for details on their age, country of residence, mental health status, a brief description of any interventions currently being undertaken (e.g., psychotherapy, CBT, EMDR), and gender. Participants will be asked if they are willing and able to engage in self-directed course content, as well as contemplative principles and practices (a brief definition of this will be offered). Participants under the age of 18, having used antipsychotic medications or recreational psychotropics, non-residents of the United Kingdom, not English speaking or diagnosed with a psychotic disorder will be thanked for their time and prevented from proceeding further with the survey. Any data gathered will be excluded from the analysis and purged.

* Participants proceeding with the study will then be asked to generate an anonymised ID code to facilitate safe handling of data storage and withdrawal.

  * Participants will then be presented with baseline assessments and provided access to Squarespace-hosted NPTS. Participants meeting inclusionary criteria will be directed to a debrief sheet (Appendix G) following the baseline assessments, reminding them of their right to withdraw and the associated process, the controls around the handling of their data, and details for local mental health organisations that they may reach out to for support should their participation have raised any concerns, including:
* Mind.org.uk - 0300 123 3393 or Email info@mind.org.uk
* Counselling-directory.org.uk - 0333 325 2500 or via their website
* Rethink Advice and Information line - 0300 5000 927

Assignment to intervention or control conditions will be set as random logic in Qualtrics.

The control group (group 2) will be on a waitlist and have access to treatment as usual (TAU), ensuring no deception, so all participants can eventually undergo the training. Following a single-blinding procedure, the TAU group will be informed that they will have access to the training (NPTS) after the end of all assessment phases (i.e., which will not take place under research conditions).

The Squarespace-hosted NPTS will remain open for a minimum of 8 weeks, during which participants in the intervention group will receive weekly email prompts reminding them to log in and engage with the content for completion of the course (once a week for 8 weeks, directly from Qualtrics).

At the post intervention 9-week mark, both groups will be prompted to retake the baseline assessments and will receive an email reminder to log in accordingly. Furthermore, a follow up assessment will be scheduled to take place 3-months after then end of the intervention, in which the same measures will be administered to the intervention and control group accordingly.

Following completion of all assessment phases, participants will receive a debrief form (Appendix H) which details the names and contact details of the researcher and supervisor and reminds participants of details for relevant mental health support resources, and thanks them for their participation. Participants will be invited to email the researcher directly should they wish to participate in a brief interview regarding their experience of NPTS. The interview schedule for the qualitative subset can be found in Appendix I. Participants will be informed that interviews will be transcribed to permit analysis for themes and feedback at a later date. This data will help to inform refinements and improvements to the program. The researcher will not video record the interview and the choice of camera on or camera off is entirely theirs.

Materials:

* Qualtrics
* Microsoft Teams
* NAS
* AAQ-II
* FFMQ
* PCL-5
* ITQ

Planned Analysis:

Within-group effects on PTSD symptoms in the Nonattachment and W/L groups will be examined using two-tailed paired samples t-tests of pre-, post and follow-up intervention scores for all measures, and within group effect sizes (Hedge's g) will be calculated. Between group effects over time will be examined using repeated-measures analyses of variance, and between group effect sizes calculated accordingly. Independent sample t-tests and chi-squared analyses will be used to examine differences between demographics and symptom measures at intake. Data will be analysed on an intention-to-treat basis.

Qualitative data will be transcribed and, through a social constructionist epistemological lens, analysed using thematic analysis following the six-phase approach:

1. Familiarisation with data

3. Searching for themes

4. Reviewing themes

5. Defining and naming themes

6. Producing the report

ELIGIBILITY:
Inclusion Criteria:

* Current or recent (within 12 months) diagnosis of PTSD (self-disclosed) OR
* Participants meeting diagnostic requirements of the ITQ OR
* Participants meeting diagnostic requirements of the PCL-C
* Participants willing and able to engage in self-directed course content (self-disclosed)
* Participants willing and able to engage with contemplative principles and practices (self-disclosed)

Exclusion Criteria:

* Non-English-speaking participants OR participants with a primary residence outside the UK
* Under the age of 18
* Participants with comorbidities such as drug or alcohol misuse which could prevent successful intervention engagement
* Participants diagnosed with a psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Nonattachment Scale | From enrollment to the end of treatment at 8 weeks, and again 3 months later.
  This study seeks to understand the impact of the program on levels of nonattachment. Details of the Nonattachment scale (NAS)can be found here: DOI: 10.1080/00223890903425960 NAS is a 30-item Likert scale informed by Buddhist principles measuring aspects such as psychological flexibility, nonreactivity, and capacity for recovery after emotional disturbance. Minimum value is 30 (all answers =1). Maximum value is 180 (all answers = 6). Higher score values are associated with better outcomes.

SECONDARY OUTCOMES:
Self-reported experiences of Post Traumatic Stress Symptoms using a combination of established trauma-based assessments, and qualitative analysis. | From enrollment to the end of treatment at 8 weeks, and again 3 months later.
  This study seeks to determine participants' experiences of trauma symptoms after accessing the intervention. The primary metric associated with assessing this outcome will be the Posttraumatic Stress Disorder 5 Checklist (PCL-5; Weathers et al., 2013) in which participants are prompted to rate on a 5-point Likert scale how much each of the 20 included problems or complaints. Higher scores indicate worse outcomes. Minimum values = 0 (20 selections of 0). Maximum values = 80 (20 selections of 4).

CONTACTS AND LOCATIONS:
Overall Officials: William Van Gordon, PhD, Study Chair — University of Derby
Locations (1):
- University of Derby, Derby, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The Research Ethics Committee of the College of Health, Psychology and Social Care at the University of Derby in accordance with the British Psychological Society (BPS) guidelines for research (2021) has reviewed and approved this study on the condition of participant anonymity. The nature of the qualitative data collected may be particularly sensitive, and there is no need to identify participants for data analysis.

REFERENCES:
- [Background] Weathers, F.W., Litz, B.T., Keane, T.M., Palmieri, P.A., Marx, B.P., & Schnurr, P.P. (2013). The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov.
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996